CLINICAL TRIAL: NCT04663646
Title: Application of Optokinetic Stimulation in the Treatment of Hemineglect
Brief Title: Optokinetic Stimulation for Hemineglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Pérez-Robledo, Fátima, Dr., University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUROUSAL02/2020
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Perceptual Disorders; Unilateral Spatial Neglect
Keywords: Perceptual Disorders; Unilateral spatial neglect; Optokinetic stimulation; Photic stimulation
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in which an intervention group will undergo optokinetic stimulation with virtual reality glasses, and the control group will receive placebo sessions.
Who Masked: Participant, Investigator
Masking Description: Participants will be assigned to one of the groups through a number contained in an opaque envelope. Only the physiotherapist in charge of applying the intervention sessions will know the assignment group of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Optokinetic stimulation
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Optokinetic stimulation — Participants are placed in a standing position, with support products, if necessary, and virtual reality glasses will be placed where the visual stimuli will be projected.
  The study will be carried out for 10 weeks with a frequency of two weekly sessions. During them, the participants will receive stimulation with OKS.
  Stimulation will be performed at 1 cm/second, the vertical black bars will move to the left. The bars change color and the participants will be asked to detect the changes that will occur in the stimulus.
  Arms: Intervention Group
Other: Placebo — Participants are placed in a standing position, with support products, if necessary, and virtual reality glasses will be placed where the visual stimuli will be projected. In this group, stimulation consists of a video with static vertical bars that change their colour at a randon intervals, in the same way that in the intervention group. The difference between groups is that in control group, bars are not in movement, preventing from generating optokinetic stimulation.
  Arms: Control Group

SUMMARY:
Hemineglect is a sequel to stroke, which appears more frequently when the injury occurs in the right cerebral hemisphere. Hemineglect refers to those patients who do not pay attention to their left side, presenting movement disorders that do not allow them to participate spontaneously in their activities of daily life.

There are different methodologies for the treatment of hemineglect. Among them, we find optokinetic stimulation (OKS), which consists of creating an illusory movement to the left to center the patient's frame of reference and thus, make them pay more attention to their left side. In recent years, the effect that this therapy has on motor movement disorders has begun to be explored, although the parameters for its correct application still seem to be unclear.

For this reason, our aim is to describe the effect that the OKS has on balance, posture, spatial representation and conscience, and movement disorders in hemineglect. Patients with hemineglect will undergo OKS to see its influence on the recovery of this sequel of stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old or older
* Diagnosis of right stroke
* Diagnosis of left heminegligence

Exclusion Criteria:

* No cooperation and comunication problems
* Uncontrolled epileptic seizures or migraines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Posture | 60 minutes
  To analyze static posture, a pressure platform will be used. It will be measured before and after the application of each experimental situation
Stability | 60 minutes
  To analyze static balance, a Carbon 5 Flex® pressure platform will be used. It will be measured before and after the application of each experimental situation
Fluff Test | 60 minutes
  It is a tool specifically designed to assess body representation in patients with hemineglect, through a body examination with closed eyes, and the removal of stickers located on both sides of the body. The percentage of stickers removed from each part of the body is assessed. It will be measured before and after the application of each experimental situation
Bisection of the line | 60 minutes
  It is one of the most used tools in the assessment of hemineglect. It consists of marking the middle of a line and evaluating how much deviation to the right occurs. The distance in centimeters to the center of the line is calculated. It will be measured before and after the application of each experimental situation
Fugl Meyer Assessment Scale | 60 minutes
  This scale assess upper limb, lower limb, balance, sensibility, range of motion and pain in patients with stroke.
Fullerton Advance Balance Test | 60 minutes
  This scale assess balance and postural control. It has a total punctuation of 40 points. People who are under 25 points have risk of fall.
Diller's cancelation test | 60 minutes
  This scale assess USN by crossing letters H included with distractors. The number of letters crossed are calculated.

SECONDARY OUTCOMES:
Sex | 1 minute
  The sex of the participants is recorded at the start of the study
Date of birth | 1 minute
  The participant's date of birth is collected in order to calculate his age in years
Date of injury | 1 minute
  The date of the injury is registered in order to calculate the time of evolution with the disease
Type of injury | 1 minute
  Description of injury to analyse if it has some effect during intervention
Admission time | 1 minute
  Date of involvement in study
National Institutes of Health Stroke Scale | 10 minutes
  is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The anonymized database (CSR) will be available from the publication of the results for 10 years in the repository of the University of Salamanca GREDOS. The study protocol, the SAP and the ICF will be published in advance.
URL: http://gredos.usal.es/

REFERENCES:
- [Derived] Perez-Robledo F, Sanchez Gonzalez JL, Bermejo-Gil BM, Llamas-Ramos R, Martin-Nogueras AM. Optokinetic stimulation effects in the management of unilateral spatial neglect in patients with chronic stroke: study protocol for a randomised controlled trial. BMJ Open. 2023 Jul 30;13(7):e070601. doi: 10.1136/bmjopen-2022-070601. PMID 37518082